CLINICAL TRIAL: NCT03976726
Title: Influence of Temperature on Volume, Weight and Density Changes of I-gel® Masks
Brief Title: Temperature Dependent Changes in I-gel Masks
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Florian Raimann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: 05/19
Record Dates: First submitted 2019-06-02; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Airway Management
Keywords: Laryngel Mask

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- i-gel size #3: Results of benchtop investigations are compared to in patient-used masks. Increasement of weight, volume expansion and decrease of density are measured.
  Interventions: Device: Comparison of physcial parameters
- i-gel size #4: Results of benchtop investigations are compared to in patient-used masks. Increasement of weight, volume expansion and decrease of density are measured.
  Interventions: Device: Comparison of physcial parameters
- i-gel size #5: Results of benchtop investigations are compared to in patient-used masks. Increasement of weight, volume expansion and decrease of density are measured.
  Interventions: Device: Comparison of physcial parameters

INTERVENTIONS:
Device: Comparison of physcial parameters — Increasement of weight, volume expansion and decrease of density are measured.

SUMMARY:
The i-gel® mask is a second generation, single use supraglottic airway device which does not have an inflatable cuff. The cuff consists of a thermoplastic elastomer and its mechanism of sealing still remains unclear. Various theories such as temperature-dependent changes in hardness and volume expansion as well as fluid absorption have been discussed.

DETAILED DESCRIPTION:
The i-gel® mask (Intersurgical, Workingham, UK), is a second generation, single use supraglottic airway device. In contrast to other devices its' cuff consists of a thermoplastic elastomer (styrene-ethylene-butadine-styrene) instead of an inflatable cuff.

Previous studies have shown, that over time the sealing improved compared to the moment of insertion. The sealing process may be based on various mechanisms. It is assumed, that the warming from room to body temperature leads to an improved adaptation to the patient-specific anatomy due to a softening of the elastomer. By definition, an elastomer is softened by the effect of temperature and become harder when reaching the glass transition temperature.

In this context, Dingley et al. described a change in the degree of hardness as a function of temperature. Prewarmed i-gel® masks (42°C, 30min.) seem to have smaller leak volumes compared to masks stored at room temperature postinsertion in paralyzed patients, but was not reproducible in non-paralyzed patients. Looking at the sealing pressure Chauhan et al. reported that i-gel® masks required a lower pressure compared to masks with an inflatable cuff.

At this point it is not yet clear, whether the thermoplastic cuff material only expands due to an increase in temperature. Liquid absorption and a consecutive expansion is also theoretically conceivable.

Therefore, the aim of the present study is to examine the i-gel® mask within the scope of a benchtop study for temperature-dependent volume expansion and liquid absorption.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery

Exclusion Criteria:

* Contraindications for the use of i-gel masks.
* Emergency operation
* non fasted patient

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Masks used in patients (n=5 per size; #3, #4, #5) requiring general anaesthesia for elective surgery without contraindications for i-gel® were collected postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Weight | Two consecutive measurements within 15 minutes once the mask temperature has cooled from body temperature to room temperature.
  Changes of masks weight.
Volume | Two consecutive measurements within 15 minutes once the mask temperature has cooled from body temperature to room temperature.
  Changes of masks volume.
Density | Two consecutive measurements within 15 minutes once the mask temperature has cooled from body temperature to room temperature.
  Changes of masks density.

CONTACTS AND LOCATIONS:
Overall Officials: Florian J Raimann, Dr., Principal Investigator — Goethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chauhan G, Nayar P, Seth A, Gupta K, Panwar M, Agrawal N. Comparison of clinical performance of the I-gel with LMA proseal. J Anaesthesiol Clin Pharmacol. 2013 Jan;29(1):56-60. doi: 10.4103/0970-9185.105798. PMID 23493414
- [Result] Gabbott DA, Beringer R. The iGEL supraglottic airway: a potential role for resuscitation? Resuscitation. 2007 Apr;73(1):161-2. doi: 10.1016/j.resuscitation.2006.10.026. Epub 2007 Feb 7. No abstract available. PMID 17289250
- [Result] Jadhav PA, Dalvi NP, Tendolkar BA. I-gel versus laryngeal mask airway-Proseal: Comparison of two supraglottic airway devices in short surgical procedures. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):221-5. doi: 10.4103/0970-9185.155153. PMID 25948905
- [Result] Janakiraman C, Chethan DB, Wilkes AR, Stacey MR, Goodwin N. A randomised crossover trial comparing the i-gel supraglottic airway and classic laryngeal mask airway. Anaesthesia. 2009 Jun;64(6):674-8. doi: 10.1111/j.1365-2044.2009.05898.x. PMID 19453322
- [Result] Russo SG, Cremer S, Eich C, Jipp M, Cohnen J, Strack M, Quintel M, Mohr A. Magnetic resonance imaging study of the in vivo position of the extraglottic airway devices i-gel and LMA-Supreme in anaesthetized human volunteers. Br J Anaesth. 2012 Dec;109(6):996-1004. doi: 10.1093/bja/aes314. Epub 2012 Sep 25. PMID 23015619
- [Result] Theiler LG, Kleine-Brueggeney M, Kaiser D, Urwyler N, Luyet C, Vogt A, Greif R, Unibe MM. Crossover comparison of the laryngeal mask supreme and the i-gel in simulated difficult airway scenario in anesthetized patients. Anesthesiology. 2009 Jul;111(1):55-62. doi: 10.1097/ALN.0b013e3181a4c6b9. PMID 19512881
- [Result] Dingley J, Stephenson J, Allender V, Dawson S, Williams D. Changes in hardness and resilience of i-gelTM cuffs with temperature: a benchtop study. Anaesthesia. 2018 Jul;73(7):856-862. doi: 10.1111/anae.14300. Epub 2018 May 3. PMID 29722434
- [Result] Komasawa N, Nishihara I, Tatsumi S, Minami T. Prewarming of the i-gel facilitates successful insertion and ventilation efficacy with muscle relaxation: a randomized study. J Clin Anesth. 2014 Dec;26(8):663-7. doi: 10.1016/j.jclinane.2014.08.009. Epub 2014 Nov 18. PMID 25468575